CLINICAL TRIAL: NCT00315757
Title: A Phase 2, Multi-Center, Open-Label, Randomized Study of Mapatumumab (TRM-1 [HGS1012], a Fully Human Monoclonal Antibody to TRAIL-R1) in Combination With Bortezomib (Velcade) and Bortezomib Alone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Mapatumumab in Combination With Bortezomib (Velcade) and Bortezomib Alone in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1012-C1055
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — mapatumumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Bortezomib
  Interventions: Drug: Bortezomib
- B-10 (Experimental): Bortezomib and Mapatumumab 10 mg/kg
  Interventions: Biological: Mapatumumab; Drug: Bortezomib
- B-20 (Experimental): Bortezomib and Mapatumumab 20 mg/kg
  Interventions: Biological: Mapatumumab; Drug: Bortezomib

INTERVENTIONS:
Biological: Mapatumumab — 10 mg/kg IV (in the vein), on day 1 of each 21-day cycle. Number of cycles: Treatment will continue for up to 17 cycles, or until disease progression or unacceptable toxicity.
  Arms: B-10
Biological: Mapatumumab — 20 mg/kg IV (in the vein), on day 1 of each 21-day cycle. Number of cycles: Treatment will continue for up to 17 cycles, or until disease progression or unacceptable toxicity.
  Arms: B-20
Drug: Bortezomib — 1.3 mg/m^2 IV (in the vein), twice weekly for two weeks (Days 1, 4, 8, and 11) of each 21-day cycle. Number of cycles: Treatment will continue for up to 17 cycles, or until disease progression or unacceptable toxicity.
  Other Names: Velcade

SUMMARY:
The purpose of this study is to evaluate the efficacy (disease response) and safety of mapatumumab in combination with bortezomib and bortezomib alone in subjects with relapsed or refractory multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple myeloma that is refractory or has relapsed after treatment
* Measurable serum and/or urine M-protein
* Failed 1 or 2 prior therapies for multiple myeloma
* 18 years of age or older

Exclusion Criteria:

* Received more than 2 prior therapies for multiple myeloma.
* Previous cancer therapies (chemotherapy, biologic therapy, radiation therapy or immunosuppressants) within the last 3 weeks
* Received monoclonal antibodies within the last 3 weeks (chimeric or murine) or 8 weeks (human or humanized)
* Received investigational (not yet approved by a regulatory authority) agent to treat multiple myeloma within the last 4 weeks
* Subjects who received a stem cell transplant using cells from themselves in the past 16 weeks
* Subjects who received a stem cell transplant using cells from another individual
* Previously treated with bortezomib or mapatumumab
* Known HIV, hepatitis-B, hepatitis-C, or hepatitis A infection
* Infection requiring antibiotics or hospitalization within the last 2 weeks
* Major surgery within the last 4 weeks
* Diagnosis with POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes)
* History of other cancers within the past 5 years
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To evaluate disease response to mapatumumab in combination with bortezomib and bortezomib alone | 17 cycles (up to a year)

SECONDARY OUTCOMES:
To evaluate the safety, including the frequency and severity of adverse events and laboratory abnormalities, of mapatumumab in combination with bortezomib and bortezomib alone throughout the study period | 17 cycles (up to a year)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Chair — GlaxoSmithKline
Locations (20):
- United States (8):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Scripps Clinic Medical Group, Inc., La Jolla, California
  - Cancer and Blood Disorders Center, Lecanto, Florida
  - University of Chicago, Chicago, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
- Australia (4):
  - Department of Haematology, Royal North Shore Hospital, St Leonards, New South Wales
  - Institute of Medical & Veterinary Science, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Clinical Haematology & BMT, Alfred Hospital, Melbourne, Victoria
- Canada (4):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Health Research Institute - General Campus, Ottawa, Ontario
  - Notre Dame Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- India (4):
  - Bharath Hospital & Institute of Oncology, Mysore, Karnataka
  - Bangalore Institute of Oncology, Bangalore
  - All India Institute of Medical Sciences, New Delhi
  - Rajiv Gandhi Cancer Institute & Research Center, New Delhi